CLINICAL TRIAL: NCT06936553
Title: Comparison of IL-8, FGF-1 and VEGF Levels in Pulpal Tissue, GCF and Dentinal Fluid Samples of Healthy, Reversible and Irreversible Pulpitis Diagnosed Teeth
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ali Erdemir, Professor doctor, Kırıkkale University
Other Study IDs: 2024/149
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-04

CONDITIONS: Pulpitis; Pulp Inflammation; Healthy Pulp; Biomarkers; Reversible Pulpitis
Keywords: pulpal diagnosis; VEGF; pulpitis; FGF-1; IL-8
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy pulp group
- Irreversible pulpitis group
- Reversible pulpitis group

SUMMARY:
This study will include 51 patients diagnosed with healthy, reversible and irreversible pulpitis. IL-8, FGF-1 and VEGF levels will be compared using pulpal tissue, gingival crevicular fluid, dentinal fluid samples collected from the teeth of these patients. First, the DOS sample will be collected non-invasively using periopaper strips without local anesthesia. Then, the caries will be cleaned by applying local anesthesia and rubber dam to the patient and a dentinal fluid sample will be collected noninvasively using PVDF membranes. In teeth with pulp exposure due to caries, the pulp tissue that needs to be removed will not be disposed of but collected as a sample. Routine root canal treatment procedures will then continue and treatment of the teeth will be completed. The collected samples will be analyzed for IL-8, FGF-1 and VEGF levels by ELISA test.

ELIGIBILITY:
Inclusion Criteria:

Control group:

* Unrestored, caries-free vital teeth with healthy pulp
* Orthodontically indicated teeth for extraction
* wisdom teeth indicated for extraction in terms of oral hygiene
* teeth that require root canal treatment for prosthetic purposes

Reversible pulpitis group:

* Teeth that react mildly to cold, hot, sour or sweet stimuli
* Teeth with no history of spontaneous pain
* Teeth that respond to cold test and electric pulp test within normal limits
* Teeth that are not sensitive to chewing or percussion

Irreversible pulpitis group:

* Teeth with a history of continuous moderate or severe spontaneous pain
* Teeth sensitive to percussion
* Teeth without periapical pathology

Exclusion Criteria:

* Patients requiring antibiotic prophylaxis.
* Patients with diabetes or haematological diseases.
* Patients who have used antibiotics or anti-inflammatory drugs in the last three weeks.
* Patients who are pregnant during treatment.
* Patients with intense plaque and tartar on their teeth, redness and bleeding in the gums.
* Patients with severe gingivitis, generalised periodontitis or periodontal pocket depth of more than 3 mm.
* Patients with no response to pulp sensitivity tests, presence of sinus tract, presence of periapical pathology on radiography.
* Teeth without pulp exposure after caries removal

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — biologically male and female patients
Study Population: The study will include patients aged between 16-60 years who presented to Kırıkkale University, Faculty of Dentistry, Department of Endodontics with the indication of root canal treatment and were diagnosed with healthy pulp status (Group 1), symptomatic irreversible pulpitis (Group 2) and asymptomatic reversible pulpitis (Group 3).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
IL-8, FGF-1 and VEGF expression levels in dentinal fluid, GCF and pulp tissue samples | Day 1
  IL-8, FGF-1 and VEGF levels will be measured in dentinal fluid, GCF and pulp tissue samples obtained during routine root canal treatment. The analysis will be performed using ELISA. The aim is to compare expression levels between patients with healthy pulp, reversible pulpitis and irreversible pulpitis.

SECONDARY OUTCOMES:
Correlation analysis between IL-8, FGF-1 and VEGF levels in dentinal fluid, GCF and pulp tissue samples | Day 1
  The study will evaluate the correlation between IL-8, FGF-1 and VEGF concentrations within and between healthy individuals, reversible pulpitis and irreversible pulpitis groups. Correlation analyses will be conducted separately for each group and comparatively between groups using appropriate statistical methods to investigate the relationships between biomarkers in pulp tissue, dentinal fluid and GCF samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University Faculty of Dentistry, Kırıkkale, Turkey (Türkiye)